CLINICAL TRIAL: NCT03786484
Title: Phase I/Ib Trial of Single Agent PBF-999 in Solid Tumour Advanced Cancer
Brief Title: Study of PBF-999 in Solid Tumour Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Palobiofarma SL (Industry)
Collaborators: Vall d'Hebron institute of oncology (VHIO), Catalan institute of oncology (Hospitalet) (ICO) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VHIO-PBF-999-01
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-01

CONDITIONS: Cancer
Keywords: solid tumors; PDE10 inhibitors; Immunoncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PBF-999 20 mg (Experimental)
  Interventions: Drug: PBF-999
- PBF-999 40 mg (Experimental)
  Interventions: Drug: PBF-999
- PBF-999 80 mg (Experimental)
  Interventions: Drug: PBF-999
- PBF-999 120 mg (Experimental)
  Interventions: Drug: PBF-999
- recommended phase 2 dose (RP2D) (Experimental)
  Interventions: Drug: PBF-999

INTERVENTIONS:
Drug: PBF-999 — Phosphodiesterase 10 inhibitor (PDE10i)

SUMMARY:
Multicentric phase I (dose escalation plus expansion) clinical trial of PBF-999 in patients with immunotherapy naïve and pretreated solid tumors to evaluate the safety, tolerability and preliminary efficacy of the compound

DETAILED DESCRIPTION:
The phase I dose escalations will be conducted utilizing the standard 3+3 dose escalation method. Pharmacokinetic (PK) data will be obtained for PBF-999.

The phase I dose expansion will consist of 1 group including immunotherapy naïve and pretreated (previous immune checkpoint inhibitors; anti-CTLA-4, anti-PD-1, anti-PD-L1 and/or combinations) solid tumors cancer patients. Pharmacodynamic (PD) data will be obtained for potential biomarker analysis with pre-treatment and on-treatment tumor biopsies.

Phase I Dose Escalation (3+3 Design):

1. The MTD will be defined as the highest dose level at which less than 2 out of 6 patients (<33%) experience DLT in Cycle 1 (first 28 days).

Phase I Safety Expansion Once RP2D has been declared for PBF-999 using the standard 3+3 design, up to 20 additional solid tumor cancer patients may be treated at the RP2D to further explore safety and tolerability of the selected PBF-999 dose.

Patients in this study will be males or females 18 years of age or older. Patients must have histologically or cytologically confirmed cancer with at least one measurable lesion, with adequate organ and marrow function, and with ECOG performance status of 0-1. Eligible patients must have received at least one prior line of therapy for their disease.

ELIGIBILITY:
Inclusion Criteria:

* Advanced/metastatic histologically confirmed solid tumor
* At least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Patients who has progressed to the standard therapy
* ECOG performance status of 0/1
* Age greater than 18 years.
* Adequate bone marrow, renal and hepatic function
* Able and willing to give valid written consent for available archival tumor samples (not mandatory) and tumor biopsies before and during protocol (immune)therapy (not mandatory but highly recommended).
* Prior immunotherapy is allowed

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 4 weeks or 5 half-lifes prior to starting on treatment.
* Symptomatic and/or untreated Brain Metastases
* Pregnancy or breast feeding
* Serious uncontrolled medical disorder or active infection that in the investigator's opinion would impair the patient's ability to receive study treatment.
* Concurrent use of other anticancer approved or investigational agents is not allowed.
* Active or prior documented autoimmune disease within the past 2 years. NOTE: Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Prior malignancy in past 2 years or as identified in Section 7.2 of this protocol
* Patients receiving systemic steroids ≥ 10mg/day of prednisone or the equivalent
* Concurrent administration of strong inhibitors or moderate inducers of CYP1A2 is not permitted; administration must be discontinued at least 7 days prior to initiating study drug administration.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 | 28 Days
  AEs will be described by system organ class and preferred tem using the Medical Dictionary for Regulatory Activities (MedDRA). Clinically relevant Laboratory abnormalities with toxicity grades according to the NCI CTCAE v4.03 will be derived and summarized.
The Maximun Tolerated Dose (MTD) of PBF-999 | 28 Days
  The MTD evaluation will be based on the Dose-limiting Toxicity (DLT) of the treated Population and will include Adverse events (AEs), Serious Adverse events (SAEs) and laboratory evaluations. DLT Evaluable Population will be all patients enrolled in the dose-escalation portion of the trial, who receive the protocol-assigned treatment with PBF-999 and complete the safety follow-up through the DLT evaluation period or experience a DLT during the DLT evaluation period.

SECONDARY OUTCOMES:
Time to PBF-999 peak concentration in plasma "Tmax | Day 1, Day 8 and Day 29
  The parameter will be calculated from plasma samples collected at days 1, day 8 and 29 after drug administration. It will consist in the time (in minutes) to reach the maximum "PBF-1129" concentration in plasma samples of patients after oral administration of PBF-999.
PBF-999 peak concentration in plasma "Cmax" | Day 1, Day 8 and Day 29
  The parameter will be calculated from plasma samples collected at days 1, 8 and 29 after drug administration. It will consist in the maximum plasma concentration (ng/mL) of PBF-999 observed after administration.
The area under PBF-999 plasma concentration-time curve to infinite time "AUC(0-inf) | Day 1, Day 8 and Day 29
  The parameter will be calculated from plasma samples collected at days 1, 8 and 29 after drug administration. It will consist in the area under the concentration-time curve from zero up to ∞ with extrapolation of the terminal phase. "AUC(0-inf)" will be given in Amount·time/ volume units
PBF-999 half-life in plasma " t½" | Day 1, Day 8 and Day 29
  The parameter will be calculated from plasma samples collected at days 1, 8 and 29 after drug administration. It will consist in the terminal half-life of PBF-999 in plasma. "t½" will be given in hours (h)
Efficacy of PBF-999 treatment as measured by Objective response rate (ORR | 2 years
  ORR: Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).ORR is defined as confirmed complete response (CR) or partial response (PR) based on modified RECIST v1.1.
Efficacy of PBF-999 as measured by Disease control rate (DCR) | 2 years
  The disease control rate (DCR) will be estimated considering the following variables: Complete response (CR), Partial response (PR) and stable disease (SD) as described by Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). These variables will be assessed based on Imaging-based evaluation methods as chest x-ray, conventional computed tomography (CT) and magnetic resonance imaging (MRI) that will be performed every 2 cycles of 28 days administration.
Efficacy of PBF-999 as measured by duration of response (DoR) | 2 years
  Duration of response (DoR) is defined as the duration from the first documentation of OR to the first documented disease progression or death due to any cause, whichever occurs first
Efficacy of PBF-999 as measured by progression-free survival (PFS) | 2 years
  Progression-free survival (PFS) will be measured from the start of treatment until the documentation of disease progression or death due to any cause, whichever occurs first. For subjects who are alive and progression-free at the time of data cut-off for analysis, PFS will be censored at the last tumor assessment date.
Efficacy of PBF-999 as measured by overall survival (OS) | 2 years
  Overall survival (OS) will be determined as the time from the start of treatment until death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Vall d'Hebron institute of oncology (VHIO), Barcelona, Spain